CLINICAL TRIAL: NCT06840756
Title: Effects of Donor-recipient Sex-matched Versus Sex-mismatched Red Blood Cell Transfusion on Outcomes in Critically Ill Adult Patients
Brief Title: Effects of Donor-recipient Sex-matched Blood Transfusion on Patient Outcomes
Acronym: SexMATTERS RCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Michelle Zeller (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Michelle Zeller, Associate Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 5080
Record Dates: First submitted 2025-01-27; First posted 2025-02-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Red Blood Cell Transfusions; Sex Differences; Health Services; Critically Ill Intensive Care Unit Patients; Hematology; Cardiovascular
Keywords: transfusions; red blood cell transfusions; sex-matched; sex-mismatched; intensive care unit; ICU; cardiovascular; circulatory; hematology; mortality; blood donor characteristics

STUDY DESIGN:
Intervention Model Description: This study is a large scale, double-blind, superiority randomized control trial (RCT).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Site blood bank and transfusion officer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sex-matched (Experimental): Sex-matched red blood cell transfusion
  Interventions: Biological: Sex-matched red blood cell transfusions
- Sex-mismatched (Active Comparator): Sex-mismatched red blood cell transfusion
  Interventions: Biological: Sex-mismatched red blood cell transfusions

INTERVENTIONS:
Biological: Sex-mismatched red blood cell transfusions — Sex-mismatched red blood cell transfusions
  Arms: Sex-mismatched
Biological: Sex-matched red blood cell transfusions — Sex-matched red blood cell transfusions
  Arms: Sex-matched

SUMMARY:
Red blood cell (RBC) transfusions are selected based upon matching donor and recipient blood group: donor and recipient sex are not considered when selecting blood for transfusion. Hence, transfused patients can currently receive sex-matched and/or unmatched RBCs when transfusions are given. Sex-matched stem cell transplants, and some solid organ transplants, have shown that sex-matching donor to recipient improves patient outcomes. Recent exploratory studies have also suggested that patient outcomes could be improved by sex-matching for RBC transfusion. There is emerging evidence of underlying biologic mechanism(s) to support these observations. This study is designed as a randomized controlled trial and will explore the impact on patients who receive RBC transfusions from donors of the same sex ("sex-matched") compared with donors of the opposite sex ("sex-mismatched").

The trial will study adult patients admitted to the Intensive Care Unit who require an RBC transfusion. Patients will be assigned (through a process called randomization) to receive sex-matched RBCs or sex-mismatched RBCs to determine if there is a difference in mortality between those receiving matched versus mismatched RBCs. The results of this trial could have direct implications on resources, blood inventory, and RBC transfusion ordering practices.

DETAILED DESCRIPTION:
Background: Red blood cell (RBC) transfusions are selected based upon donor and recipient blood group compatibility without consideration of donor and recipient sex. Stem cell transplants, and some solid organ transplants, have shown that sex-matching donor to recipient improves patient outcomes. The Principal Investigator has completed a systematic review/meta-analysis and a 40,000 patient exploratory analysis; both showed a signal of benefit from sex-matched RBC transfusion. Biological findings to support the hypothesis that sex-matched RBC transfusions improve survival in recipients are also emerging.

Controversial results have emerged from observational studies and a randomized controlled trial (RCT) regarding recipient mortality from sex-mismatched RBC transfusions; hence, equipoise exists.

The Principal Investigator completed a multisite pilot RCT that showed feasibility for conducting a large-scale RCT and has helped to inform design for this study proposal. The goal of this research project is to develop a precision transfusion strategy based on sex-matching of blood donor and recipient to minimize adverse effects and improve patient outcomes post-transfusion.

Overall Research Question: In transfused adult patients admitted to the Intensive Care Unit (ICU), do donor-recipient sex-matched RBC transfusions result in improved mortality compared to sex-mismatched RBC transfusions?

Methods: This study is a superiority RCT with pragmatic features that will occur across participating sites in Canada.

Study population: adult patients (age≥18) who are hospitalized with admission to an eligible ICU and requiring RBC transfusion.

Intervention: donor-recipient sex-matched RBC transfusions. Comparison: donor-recipient sex-mismatched RBC transfusions.

Primary Outcome: 30 day mortality from time of randomization. Secondary Outcomes: time to death, 30 day in-hospital mortality, 90 day mortality, hemoglobin and creatinine increment, ICU and hospital lengths of stay, number/type of transfused products and cost effectiveness analysis. Subgroup analyses will consider recipient sex, age, transfusion exposure, blood type, admitting diagnosis, baseline hemoglobin/creatinine.

Expertise: The study team is uniquely positioned with extensive knowledge and expertise in transfusion medicine, research methodology, conduct of large pragmatic trials, and biostatistics. The study team will collaborate with Canadian Blood Services and experts in blood utilization, and operational modeling. This study is supported and endorsed by the Canadian Transfusion Trials Group.

Importance & Outcomes: Anemia is common in critically ill patients; as many as 90% of patients will become anemic by the third day of their ICU admission. Between 20% and 40% of critically ill patients admitted to the ICU will require RBC transfusion; each patient will receive on average 2 to 5 RBC units. The Age of Blood Evaluation (ABLE) study showed a 90 day all cause mortality rate of 35-37% in the transfused ICU population studied. The pilot study reflected similar mortality rates. If providing sex-matched transfusions can decrease mortality, this could translate to high numbers of preventable deaths given that 85 million RBC units are transfused globally each year. If this study finds that donor-recipient sex-matching saves lives, this would require changes at the level of the blood supplier to identify sex on each RBC unit, and changes at the hospital level that would incorporate sex-matching into the selection of compatible blood for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18);
* Admission to a participating ICU;
* Requiring RBC transfusion.

Exclusion Criteria:

* Requirement for a specialized RBC product or unit not readily available in inventory (e.g., rare blood type, washed RBCs, complex RBC antibodies, etc.);
* Massively bleeding patient (i.e., ≥4 units of blood ordered at one time, or Massive Hemorrhage Protocol initiated, or an urgent blood request made);
* Sex unknown or sex other than male or female (i.e. intersex);
* Do not have a valid Ontario Health Insurance Plan (OHIP) health card number.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11082 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
30 day mortality | From randomization to 30 days post-randomization.
  Death within 30 days of randomization.

SECONDARY OUTCOMES:
30 day in-hospital mortality | From randomization to 30 days post-randomization.
  In-hospital death within 30 days of randomization.
90 day mortality | From randomization to 90 days post-randomization.
  Death within 90 days of randomization.
Time to 30 day in-hospital mortality | From randomization to 30 days post-randomization.
  Time to in-hospital death within 30 days of randomization.
Hemoglobin increment | From time of randomization until death or discharge from ICU; up to 90 days post randomization.
  Lowest hemoglobin post-randomization during ICU admission.
Need for renal replacement therapy | From time of randomization during ICU admission, until death or discharge from ICU; up to 90 days post randomization.
  Need for renal replacement therapy e.g. CRRT or HD post randomization during ICU admission.
ICU/hospital length of stay | From randomization to 30 days post-randomization.
  The number of ICU-free days over 30 days and the number of days in hospital over 30 days.
Number/type/volume/dose of transfused product | From randomization to 90 days post-randomization.
  Total number of transfusion interventions, cumulative proportion of units received that were from a sex-mismatched donor
Transfusion reactions | From randomization to 30 days post-randomization.
  Reactions related to RBC transfusions.
Cost effectiveness | From randomization to 90 days post-randomization.
  Cost effectiveness measured using the incremental cost per life year saved (ICER) between sex-matched and mismatched transfusions.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Zeller, Doctor of Medicine, Principal Investigator — McMaster University
Locations (8):
- Canada (8):
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared.

REFERENCES:
- [Background] Alshalani A, van Manen L, Boshuizen M, van Bruggen R, Acker JP, Juffermans NP. The Effect of Sex-Mismatched Red Blood Cell Transfusion on Endothelial Cell Activation in Critically Ill Patients. Transfus Med Hemother. 2021 Nov 24;49(2):98-105. doi: 10.1159/000520651. eCollection 2022 Apr. PMID 35611381
- [Background] Aubron C, Nichol A, Cooper DJ, Bellomo R. Age of red blood cells and transfusion in critically ill patients. Ann Intensive Care. 2013 Jan 15;3(1):2. doi: 10.1186/2110-5820-3-2. PMID 23316800
- [Background] Zeller MP, Barty R, Aandahl A, Apelseth TO, Callum J, Dunbar NM, Elahie A, Garritsen H, Hancock H, Kutner JM, Manukian B, Mizuta S, Okuda M, Pagano MB, Poglod R, Rushford K, Selleng K, Sorensen CH, Sprogoe U, Staves J, Weiland T, Wendel S, Wood EM, van de Watering L, van Wordragen-Vlaswinkel M, Ziman A, Jan Zwaginga J, Murphy MF, Heddle NM, Yazer MH; Biomedical Excellence for Safer Transfusion (BEST) Collaborative. An international investigation into O red blood cell unit administration in hospitals: the GRoup O Utilization Patterns (GROUP) study. Transfusion. 2017 Oct;57(10):2329-2337. doi: 10.1111/trf.14255. Epub 2017 Aug 25. PMID 28840943
- [Background] Zeller MP, Barty R, Dunbar NM, Elahie A, Flanagan P, Garritsen H, Kutner JM, Pagano MB, Poglod R, Rogers TS, Staves J, van Wordragen-Vlaswinkel M, Zwaginga JJ, Murphy MF, Heddle NM, Yazer MH; Biomedical Excellence for Safer Transfusion (BEST) Collaborative. An international investigation into AB plasma administration in hospitals: how many AB plasma units were infused? The HABSWIN study. Transfusion. 2018 Jan;58(1):151-157. doi: 10.1111/trf.14368. Epub 2017 Oct 14. PMID 29030954
- [Background] Friede T, Kieser M. Blinded sample size re-estimation in superiority and noninferiority trials: bias versus variance in variance estimation. Pharm Stat. 2013 May-Jun;12(3):141-6. doi: 10.1002/pst.1564. Epub 2013 Mar 19. PMID 23509095
- [Background] Leach Bennett J, Blajchman MA, Delage G, Fearon M, Devine D. Proceedings of a consensus conference: Risk-Based Decision Making for Blood Safety. Transfus Med Rev. 2011 Oct;25(4):267-92. doi: 10.1016/j.tmrv.2011.05.002. Epub 2011 Jul 16. PMID 21763103
- [Background] Cooper DJ, McQuilten ZK, Nichol A, Ady B, Aubron C, Bailey M, Bellomo R, Gantner D, Irving DO, Kaukonen KM, McArthur C, Murray L, Pettila V, French C; TRANSFUSE Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Age of Red Cells for Transfusion and Outcomes in Critically Ill Adults. N Engl J Med. 2017 Nov 9;377(19):1858-1867. doi: 10.1056/NEJMoa1707572. Epub 2017 Sep 27. PMID 28952891
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908
- [Background] Asfar P, Meziani F, Hamel JF, Grelon F, Megarbane B, Anguel N, Mira JP, Dequin PF, Gergaud S, Weiss N, Legay F, Le Tulzo Y, Conrad M, Robert R, Gonzalez F, Guitton C, Tamion F, Tonnelier JM, Guezennec P, Van Der Linden T, Vieillard-Baron A, Mariotte E, Pradel G, Lesieur O, Ricard JD, Herve F, du Cheyron D, Guerin C, Mercat A, Teboul JL, Radermacher P; SEPSISPAM Investigators. High versus low blood-pressure target in patients with septic shock. N Engl J Med. 2014 Apr 24;370(17):1583-93. doi: 10.1056/NEJMoa1312173. Epub 2014 Mar 18. PMID 24635770
- [Background] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363
- [Background] Barrot L, Asfar P, Mauny F, Winiszewski H, Montini F, Badie J, Quenot JP, Pili-Floury S, Bouhemad B, Louis G, Souweine B, Collange O, Pottecher J, Levy B, Puyraveau M, Vettoretti L, Constantin JM, Capellier G; LOCO2 Investigators and REVA Research Network. Liberal or Conservative Oxygen Therapy for Acute Respiratory Distress Syndrome. N Engl J Med. 2020 Mar 12;382(11):999-1008. doi: 10.1056/NEJMoa1916431. PMID 32160661
- [Background] Rochwerg B, Millen T, Austin P, Zeller M, D'Aragon F, Jaeschke R, Masse MH, Mehta S, Lamontagne F, Meade M, Guyatt G, Cook DJ; Canadian Critical Care Trials Group. Fluids in Sepsis and Septic Shock (FISSH): protocol for a pilot randomised controlled trial. BMJ Open. 2017 Jul 20;7(7):e017602. doi: 10.1136/bmjopen-2017-017602. PMID 28729329
- [Background] Friedrich JO, Harhay MO, Angus DC, Burns KEA, Cook DJ, Fergusson DA, Finfer S, Hebert P, Rowan K, Rubenfeld G, Marshall JC; International Forum for Acute Care Trialists (InFACT). Mortality As a Measure of Treatment Effect in Clinical Trials Recruiting Critically Ill Patients. Crit Care Med. 2023 Feb 1;51(2):222-230. doi: 10.1097/CCM.0000000000005721. Epub 2023 Jan 20. PMID 36661450
- [Background] Heddle NM, Cook RJ, Arnold DM, Liu Y, Barty R, Crowther MA, Devereaux PJ, Hirsh J, Warkentin TE, Webert KE, Roxby D, Sobieraj-Teague M, Kurz A, Sessler DI, Figueroa P, Ellis M, Eikelboom JW. Effect of Short-Term vs. Long-Term Blood Storage on Mortality after Transfusion. N Engl J Med. 2016 Nov 17;375(20):1937-1945. doi: 10.1056/NEJMoa1609014. Epub 2016 Oct 24. PMID 27775503
- [Background] Chasse M, Fergusson DA, Tinmouth A, Acker JP, Perelman I, Tuttle A, English SW, Hawken S, Forster AJ, Shehata N, Thavorn K, Wilson K, Cober N, Maddison H, Tokessy M. Effect of Donor Sex on Recipient Mortality in Transfusion. N Engl J Med. 2023 Apr 13;388(15):1386-1395. doi: 10.1056/NEJMoa2211523. PMID 37043654
- [Background] Schandelmaier S, Briel M, Varadhan R, Schmid CH, Devasenapathy N, Hayward RA, Gagnier J, Borenstein M, van der Heijden GJMG, Dahabreh IJ, Sun X, Sauerbrei W, Walsh M, Ioannidis JPA, Thabane L, Guyatt GH. Development of the Instrument to assess the Credibility of Effect Modification Analyses (ICEMAN) in randomized controlled trials and meta-analyses. CMAJ. 2020 Aug 10;192(32):E901-E906. doi: 10.1503/cmaj.200077. PMID 32778601
- [Background] Alshalani A, de Wissel MB, Tuip-de Boer AM, Roelofs JJTH, van Bruggen R, Acker JP, Juffermans NP. Transfusion of female blood in a rat model is associated with red blood cells entrapment in organs. PLoS One. 2023 Nov 22;18(11):e0288308. doi: 10.1371/journal.pone.0288308. eCollection 2023. PMID 37992035
- [Background] Elahi S. New insight into an old concept: role of immature erythroid cells in immune pathogenesis of neonatal infection. Front Immunol. 2014 Aug 12;5:376. doi: 10.3389/fimmu.2014.00376. eCollection 2014. PMID 25161654
- [Background] Gutierrez M, Fish MB, Golinski AW, Eniola-Adefeso O. Presence of Rigid Red Blood Cells in Blood Flow Interferes with the Vascular Wall Adhesion of Leukocytes. Langmuir. 2018 Feb 13;34(6):2363-2372. doi: 10.1021/acs.langmuir.7b03890. Epub 2018 Jan 31. PMID 29347819
- [Background] Li W, Acker JP. Immunological impact of the CD71+ RBCs: A potential immune mediator in transfusion. Transfus Apher Sci. 2023 Jun;62(3):103721. doi: 10.1016/j.transci.2023.103721. Epub 2023 May 8. PMID 37173208
- [Background] Chan KT, Choi MY, Lai KK, Tan W, Tung LN, Lam HY, Tong DK, Lee NP, Law S. Overexpression of transferrin receptor CD71 and its tumorigenic properties in esophageal squamous cell carcinoma. Oncol Rep. 2014 Mar;31(3):1296-304. doi: 10.3892/or.2014.2981. Epub 2014 Jan 16. PMID 24435655
- [Background] Liu Q, Wang M, Hu Y, Xing H, Chen X, Zhang Y, Zhu P. Significance of CD71 expression by flow cytometry in diagnosis of acute leukemia. Leuk Lymphoma. 2014 Apr;55(4):892-8. doi: 10.3109/10428194.2013.819100. Epub 2013 Aug 20. PMID 23962073
- [Background] Miller D, Romero R, Unkel R, Xu Y, Vadillo-Ortega F, Hassan SS, Gomez-Lopez N. CD71+ erythroid cells from neonates born to women with preterm labor regulate cytokine and cellular responses. J Leukoc Biol. 2018 Apr;103(4):761-775. doi: 10.1002/JLB.5A0717-291RRR. Epub 2018 Feb 1. PMID 29389020
- [Background] Namdar A, Koleva P, Shahbaz S, Strom S, Gerdts V, Elahi S. CD71+ erythroid suppressor cells impair adaptive immunity against Bordetella pertussis. Sci Rep. 2017 Aug 10;7(1):7728. doi: 10.1038/s41598-017-07938-7. PMID 28798335
- [Background] Elahi S, Ertelt JM, Kinder JM, Jiang TT, Zhang X, Xin L, Chaturvedi V, Strong BS, Qualls JE, Steinbrecher KA, Kalfa TA, Shaaban AF, Way SS. Immunosuppressive CD71+ erythroid cells compromise neonatal host defence against infection. Nature. 2013 Dec 5;504(7478):158-62. doi: 10.1038/nature12675. Epub 2013 Nov 6. PMID 24196717
- [Background] Li W, William N, Acker JP. Donor sex, pre-donation hemoglobin, and manufacturing affect CD71+ cells in red cell concentrates. Transfusion. 2023 Mar;63(3):601-609. doi: 10.1111/trf.17250. Epub 2023 Jan 19. PMID 36655728
- [Background] Gladwin MT, Kanias T, Kim-Shapiro DB. Hemolysis and cell-free hemoglobin drive an intrinsic mechanism for human disease. J Clin Invest. 2012 Apr;122(4):1205-8. doi: 10.1172/JCI62972. Epub 2012 Mar 26. PMID 22446184
- [Background] Hod EA, Spitalnik SL. Stored red blood cell transfusions: Iron, inflammation, immunity, and infection. Transfus Clin Biol. 2012 Jun;19(3):84-9. doi: 10.1016/j.tracli.2012.04.001. Epub 2012 Jun 7. PMID 22682673
- [Background] Donadee C, Raat NJ, Kanias T, Tejero J, Lee JS, Kelley EE, Zhao X, Liu C, Reynolds H, Azarov I, Frizzell S, Meyer EM, Donnenberg AD, Qu L, Triulzi D, Kim-Shapiro DB, Gladwin MT. Nitric oxide scavenging by red blood cell microparticles and cell-free hemoglobin as a mechanism for the red cell storage lesion. Circulation. 2011 Jul 26;124(4):465-76. doi: 10.1161/CIRCULATIONAHA.110.008698. Epub 2011 Jul 11. PMID 21747051
- [Background] Roubinian NH, Plimier C, Woo JP, Lee C, Bruhn R, Liu VX, Escobar GJ, Kleinman SH, Triulzi DJ, Murphy EL, Busch MP. Effect of donor, component, and recipient characteristics on hemoglobin increments following red blood cell transfusion. Blood. 2019 Sep 26;134(13):1003-1013. doi: 10.1182/blood.2019000773. Epub 2019 Jul 26. PMID 31350268
- [Background] Minneci PC, Deans KJ, Zhi H, Yuen PS, Star RA, Banks SM, Schechter AN, Natanson C, Gladwin MT, Solomon SB. Hemolysis-associated endothelial dysfunction mediated by accelerated NO inactivation by decompartmentalized oxyhemoglobin. J Clin Invest. 2005 Dec;115(12):3409-17. doi: 10.1172/JCI25040. Epub 2005 Nov 17. PMID 16294219
- [Background] William N, Osmani R, Acker JP. Towards the crux of sex-dependent variability in red cell concentrates. Transfus Apher Sci. 2023 Dec;62(6):103827. doi: 10.1016/j.transci.2023.103827. Epub 2023 Sep 29. PMID 37793959
- [Background] Alshalani A, Li W, Juffermans NP, Seghatchian J, Acker JP. Biological mechanisms implicated in adverse outcomes of sex mismatched transfusions. Transfus Apher Sci. 2019 Jun;58(3):351-356. doi: 10.1016/j.transci.2019.04.023. Epub 2019 May 1. PMID 31064732
- [Background] Tzounakas VL, Kriebardis AG, Papassideri IS, Antonelou MH. Donor-variation effect on red blood cell storage lesion: A close relationship emerges. Proteomics Clin Appl. 2016 Aug;10(8):791-804. doi: 10.1002/prca.201500128. Epub 2016 May 23. PMID 27095294
- [Background] Kameneva MV, Watach MJ, Borovetz HS. Gender difference in rheologic properties of blood and risk of cardiovascular diseases. Clin Hemorheol Microcirc. 1999;21(3-4):357-63. PMID 10711771
- [Background] Kanias T, Lanteri MC, Page GP, Guo Y, Endres SM, Stone M, Keating S, Mast AE, Cable RG, Triulzi DJ, Kiss JE, Murphy EL, Kleinman S, Busch MP, Gladwin MT. Ethnicity, sex, and age are determinants of red blood cell storage and stress hemolysis: results of the REDS-III RBC-Omics study. Blood Adv. 2017 Jun 27;1(15):1132-1141. doi: 10.1182/bloodadvances.2017004820. PMID 29034365
- [Background] Lanteri MC, Kanias T, Keating S, Stone M, Guo Y, Page GP, Brambilla DJ, Endres-Dighe SM, Mast AE, Bialkowski W, D'Andrea P, Cable RG, Spencer BR, Triulzi DJ, Murphy EL, Kleinman S, Gladwin MT, Busch MP; NHLBI Recipient Epidemiology Donor Evaluation Study (REDS)-III Program. Intradonor reproducibility and changes in hemolytic variables during red blood cell storage: results of recall phase of the REDS-III RBC-Omics study. Transfusion. 2019 Jan;59(1):79-88. doi: 10.1111/trf.14987. Epub 2018 Nov 8. PMID 30408207
- [Background] Jordan A, Chen D, Yi QL, Kanias T, Gladwin MT, Acker JP. Assessing the influence of component processing and donor characteristics on quality of red cell concentrates using quality control data. Vox Sang. 2016 Jul;111(1):8-15. doi: 10.1111/vox.12378. Epub 2016 Mar 18. PMID 26991891
- [Background] Kanias T, Sinchar D, Osei-Hwedieh D, Baust JJ, Jordan A, Zimring JC, Waterman HR, de Wolski KS, Acker JP, Gladwin MT. Testosterone-dependent sex differences in red blood cell hemolysis in storage, stress, and disease. Transfusion. 2016 Oct;56(10):2571-2583. doi: 10.1111/trf.13745. Epub 2016 Aug 9. PMID 27507802
- [Background] Fergusson DA, Chasse M, Tinmouth A, Acker JP, English S, Forster AJ, Hawken S, Shehata N, Thavorn K, Wilson K, Tuttle A, Perelman I, Cober N, Maddison H, Tokessy M. Pragmatic, double-blind, randomised trial evaluating the impact of red blood cell donor sex on recipient mortality in an academic hospital population: the innovative Trial Assessing Donor Sex (iTADS) protocol. BMJ Open. 2021 Feb 23;11(2):e049598. doi: 10.1136/bmjopen-2021-049598. PMID 33622960
- [Background] Alshalani A, Uhel F, Cremer OL, Schultz MJ, de Vooght KMK, van Bruggen R, Acker JP, Juffermans NP. Donor-recipient sex is associated with transfusion-related outcomes in critically ill patients. Blood Adv. 2022 Jun 14;6(11):3260-3267. doi: 10.1182/bloodadvances.2021006402. PMID 35286383
- [Background] Edgren G, Murphy EL, Brambilla DJ, Westlake M, Rostgaard K, Lee C, Cable RG, Triulzi D, Bruhn R, St Lezin EM, Erikstrup C, Ullum H, Glynn SA, Kleinman S, Hjalgrim H, Roubinian NH; NHLBI Recipient Epidemiology and Donor Evaluation Study-III (REDS-III) Group. Association of Blood Donor Sex and Prior Pregnancy With Mortality Among Red Blood Cell Transfusion Recipients. JAMA. 2019 Jun 11;321(22):2183-2192. doi: 10.1001/jama.2019.7084. PMID 31184739
- [Background] Patel RM, Lukemire J, Shenvi N, Arthur C, Stowell SR, Sola-Visner M, Easley K, Roback JD, Guo Y, Josephson CD. Association of Blood Donor Sex and Age With Outcomes in Very Low-Birth-Weight Infants Receiving Blood Transfusion. JAMA Netw Open. 2021 Sep 1;4(9):e2123942. doi: 10.1001/jamanetworkopen.2021.23942. PMID 34477851
- [Background] Bahr TM, Christensen TR, Tweddell SM, Henry E, Rees T, Astin ME, Kelley WE, Ilstrup SJ, Ohls RK, Christensen RD. Associations between blood donor sex and age, and outcomes of transfused newborn infants. Transfusion. 2023 Jul;63(7):1290-1297. doi: 10.1111/trf.17417. Epub 2023 May 22. PMID 37218104
- [Background] Holzmann MJ, Sartipy U, Olsson ML, Dickman P, Edgren G. Sex-Discordant Blood Transfusions and Survival After Cardiac Surgery: A Nationwide Cohort Study. Circulation. 2016 Nov 22;134(21):1692-1694. doi: 10.1161/CIRCULATIONAHA.116.025087. No abstract available. PMID 27881511
- [Background] Desmarets M, Bardiaux L, Benzenine E, Dussaucy A, Binda D, Tiberghien P, Quantin C, Monnet E. Effect of storage time and donor sex of transfused red blood cells on 1-year survival in patients undergoing cardiac surgery: an observational study. Transfusion. 2016 May;56(5):1213-22. doi: 10.1111/trf.13537. Epub 2016 Mar 2. PMID 26935140
- [Background] Bjursten H, Dardashti A, Bjork J, Wierup P, Algotsson L, Ederoth P. Transfusion of sex-mismatched and non-leukocyte-depleted red blood cells in cardiac surgery increases mortality. J Thorac Cardiovasc Surg. 2016 Jul;152(1):223-232.e1. doi: 10.1016/j.jtcvs.2015.12.022. Epub 2015 Dec 19. PMID 26874600
- [Background] Middelburg RA, Briet E, van der Bom JG. Mortality after transfusions, relation to donor sex. Vox Sang. 2011 Oct;101(3):221-9. doi: 10.1111/j.1423-0410.2011.01487.x. Epub 2011 Apr 8. PMID 21477152
- [Background] Zeller MP, Rochwerg B, Jamula E, Li N, Hillis C, Acker JP, Runciman RJR, Lane SJ, Ahmed N, Arnold DM, Heddle NM. Sex-mismatched red blood cell transfusions and mortality: A systematic review and meta-analysis. Vox Sang. 2019 Jul;114(5):505-516. doi: 10.1111/vox.12783. Epub 2019 May 23. PMID 31124172
- [Background] Heddle NM, Cook RJ, Liu Y, Zeller M, Barty R, Acker JP, Eikelboom J, Arnold DM. The association between blood donor sex and age and transfusion recipient mortality: an exploratory analysis. Transfusion. 2019 Feb;59(2):482-491. doi: 10.1111/trf.15011. Epub 2018 Nov 10. PMID 30414291
- [Background] Lacroix J, Hebert PC, Fergusson DA, Tinmouth A, Cook DJ, Marshall JC, Clayton L, McIntyre L, Callum J, Turgeon AF, Blajchman MA, Walsh TS, Stanworth SJ, Campbell H, Capellier G, Tiberghien P, Bardiaux L, van de Watering L, van der Meer NJ, Sabri E, Vo D; ABLE Investigators; Canadian Critical Care Trials Group. Age of transfused blood in critically ill adults. N Engl J Med. 2015 Apr 9;372(15):1410-8. doi: 10.1056/NEJMoa1500704. Epub 2015 Mar 17. PMID 25853745
- [Background] Kollman C, Howe CW, Anasetti C, Antin JH, Davies SM, Filipovich AH, Hegland J, Kamani N, Kernan NA, King R, Ratanatharathorn V, Weisdorf D, Confer DL. Donor characteristics as risk factors in recipients after transplantation of bone marrow from unrelated donors: the effect of donor age. Blood. 2001 Oct 1;98(7):2043-51. doi: 10.1182/blood.v98.7.2043. PMID 11567988
- [Background] Jagasia M, Arora M, Flowers ME, Chao NJ, McCarthy PL, Cutler CS, Urbano-Ispizua A, Pavletic SZ, Haagenson MD, Zhang MJ, Antin JH, Bolwell BJ, Bredeson C, Cahn JY, Cairo M, Gale RP, Gupta V, Lee SJ, Litzow M, Weisdorf DJ, Horowitz MM, Hahn T. Risk factors for acute GVHD and survival after hematopoietic cell transplantation. Blood. 2012 Jan 5;119(1):296-307. doi: 10.1182/blood-2011-06-364265. Epub 2011 Oct 18. PMID 22010102
- [Background] Nannya Y, Kataoka K, Hangaishi A, Imai Y, Takahashi T, Kurokawa M. The negative impact of female donor/male recipient combination in allogeneic hematopoietic stem cell transplantation depends on disease risk. Transpl Int. 2011 May;24(5):469-76. doi: 10.1111/j.1432-2277.2011.01229.x. Epub 2011 Feb 5. PMID 21294789
- [Background] Nakasone H, Remberger M, Tian L, Brodin P, Sahaf B, Wu F, Mattsson J, Lowsky R, Negrin R, Miklos DB, Meyer E. Risks and benefits of sex-mismatched hematopoietic cell transplantation differ according to conditioning strategy. Haematologica. 2015 Nov;100(11):1477-85. doi: 10.3324/haematol.2015.125294. Epub 2015 Aug 6. PMID 26250581
- [Background] Khush KK, Kubo JT, Desai M. Influence of donor and recipient sex mismatch on heart transplant outcomes: analysis of the International Society for Heart and Lung Transplantation Registry. J Heart Lung Transplant. 2012 May;31(5):459-66. doi: 10.1016/j.healun.2012.02.005. Epub 2012 Mar 13. PMID 22418079
- [Background] Weiss ES, Allen JG, Patel ND, Russell SD, Baumgartner WA, Shah AS, Conte JV. The impact of donor-recipient sex matching on survival after orthotopic heart transplantation: analysis of 18 000 transplants in the modern era. Circ Heart Fail. 2009 Sep;2(5):401-8. doi: 10.1161/CIRCHEARTFAILURE.108.844183. Epub 2009 Jul 8. PMID 19808369
- [Background] Stern M, Passweg JR, Locasciulli A, Socie G, Schrezenmeier H, Bekassy AN, Fuehrer M, Hows J, Korthof ET, McCann S, Tichelli A, Zoumbos NC, Marsh JC, Bacigalupo A, Gratwohl A; Aplastic Anemia Working Party of the European Group for Blood and Marrow Transplantation. Influence of donor/recipient sex matching on outcome of allogeneic hematopoietic stem cell transplantation for aplastic anemia. Transplantation. 2006 Jul 27;82(2):218-26. doi: 10.1097/01.tp.0000226156.99206.d1. PMID 16858285
- [Background] Lin Y, Saw CL, Hannach B, Goldman M. Transfusion-related acute lung injury prevention measures and their impact at Canadian Blood Services. Transfusion. 2012 Mar;52(3):567-74. doi: 10.1111/j.1537-2995.2011.03330.x. Epub 2011 Sep 2. PMID 21895676
- [Background] Lieberman L, Petraszko T, Yi QL, Hannach B, Skeate R. Transfusion-related lung injury in children: a case series and review of the literature. Transfusion. 2014 Jan;54(1):57-64. doi: 10.1111/trf.12249. Epub 2013 Jun 13. PMID 23763359
- [Background] Caram-Deelder C, Kreuger AL, Evers D, de Vooght KMK, van de Kerkhof D, Visser O, Pequeriaux NCV, Hudig F, Zwaginga JJ, van der Bom JG, Middelburg RA. Association of Blood Transfusion From Female Donors With and Without a History of Pregnancy With Mortality Among Male and Female Transfusion Recipients. JAMA. 2017 Oct 17;318(15):1471-1478. doi: 10.1001/jama.2017.14825. PMID 29049654
- [Background] Edgren G, Ullum H, Rostgaard K, Erikstrup C, Sartipy U, Holzmann MJ, Nyren O, Hjalgrim H. Association of Donor Age and Sex With Survival of Patients Receiving Transfusions. JAMA Intern Med. 2017 Jun 1;177(6):854-860. doi: 10.1001/jamainternmed.2017.0890. PMID 28437543
- [Background] Chasse M, Tinmouth A, English SW, Acker JP, Wilson K, Knoll G, Shehata N, van Walraven C, Forster AJ, Ramsay T, McIntyre LA, Fergusson DA. Association of Blood Donor Age and Sex With Recipient Survival After Red Blood Cell Transfusion. JAMA Intern Med. 2016 Sep 1;176(9):1307-14. doi: 10.1001/jamainternmed.2016.3324. PMID 27398639
- [Background] Carson JL, Grossman BJ, Kleinman S, Tinmouth AT, Marques MB, Fung MK, Holcomb JB, Illoh O, Kaplan LJ, Katz LM, Rao SV, Roback JD, Shander A, Tobian AA, Weinstein R, Swinton McLaughlin LG, Djulbegovic B; Clinical Transfusion Medicine Committee of the AABB. Red blood cell transfusion: a clinical practice guideline from the AABB*. Ann Intern Med. 2012 Jul 3;157(1):49-58. doi: 10.7326/0003-4819-157-1-201206190-00429. PMID 22751760
- [Background] Pfuntner A, Wier LM, Stocks C. Most Frequent Procedures Performed in U.S. Hospitals, 2011. 2013 Oct. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #165. Available from http://www.ncbi.nlm.nih.gov/books/NBK174682/ PMID 24354027
- See also: American Red Cross: Blood Facts and Statistics — http://www.redcrossblood.org/learn-about-blood/blood-facts-and-statistics
- See also: Mykhailova O, Li W, Acker JP. RBC subpopulations in stored concentrates have different quality characteristics. Transfusion. 2019;59(S3):81A — https://aabb.confex.com/aabb/2019/meetingapp.cgi/Paper/6901
- See also: Tri-Council Policy Statement. Ethical Conduct for Research Involving Humans TCPS2. Vol 45.; 2022 — https://ethics.gc.ca/eng/policy-politique_tcps2-eptc2_2022.html
- See also: Iron K, Zagorski B, Sykora K, Manuel D. Living and Dying in Ontario : An Opportunity for Improved Health Information; ICES Investigative Report.; 2008 — https://www.ices.on.ca/wp-content/uploads/2023/06/Full-report-21.pdf
- See also: Therneau T, Grambsch P. Modeling Survival Data: Extending the Cox Model. New York, NY: Springer-Verlag; 2000 — https://doi.org/10.1007/978-1-4757-3294-8
- See also: 1. Zeller M, Cook R, Arnold D, et al. Sex-Matched Compared to Sex-Mismatched Red Blood Cell Transfusion: A Pilot Randomized Controlled Trial. In: Canadian Society for Transfusion Medicine Annual Meeting. Montreal; 2023:Oral Abstract Presentation — https://www.researchgate.net/publication/380151180_Sex-matched_compared_to_sex-mismatched_red_blood_cell_transfusion_a_pilot_randomized_controlled_trial

DOCUMENTS (1):
  • Study Protocol (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT06840756/Prot_001.pdf